CLINICAL TRIAL: NCT01012479
Title: Clinical Study to Evaluate the Efficacy and Safety of the Combination Therapy Candesartan Cilexetil 32 mg Plus Hydrochlorothiazide 25 mg in Patients With Severe Hypertension
Brief Title: Efficacy and Safety of Candesartan Cilexetil Plus Hydrochlorothiazide in Subjects With Severe Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Medical Director, Takeda Pharma GmbH, Aachen (Germany)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLO K027; DE-CAN-027 (Other: Takeda ID); 2009-011776-30 (EudraCT Number); U1111-1112-2376 (Registry Identifier: WHO)
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-07

CONDITIONS: Hypertension
Keywords: Blood Pressure; Blood Pressure, High; Drug Therapy
MeSH Terms: conditions — Hypertension | interventions — candesartan cilexetil; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Candesartan QD + Hydrochlorothiazide QD (Experimental)
  Interventions: Drug: Candesartan cilexetil and hydrochlorothiazide

INTERVENTIONS:
Drug: Candesartan cilexetil and hydrochlorothiazide — Candesartan cilexetil 16 mg, tablets, orally, once daily for 1 week; increased to candesartan cilexetil 16 mg and hydrochlorothiazide 12.5 mg combination tablet, orally once daily for 2 weeks; then increased to candesartan cilexetil 32 mg and hydrochlorothiazide 25 mg combination tablets, orally, once daily for up to 6 weeks
  Other Names: Blopress; Atacand®; Amias; Ratacand; Kenzen; Blopressid

SUMMARY:
The purpose of this study is to see if Candesartan, once daily (QD), added with Hydrochlorothiazide may be helpful in treating people with newly diagnosed severe essential hypertension.

DETAILED DESCRIPTION:
Medical data show a link between blood pressure and the risk of heart disease (cardiovascular disease) such as stroke and heart attack. Clinical trials have shown that lowering blood pressure in patients with high blood pressure (hypertension) reduces the number of cardiovascular events.

Many people still have untreated hypertension. There are many reasons why target blood pressure is not reached. One is that most patients need more than one antihypertensive drug in order to lower high blood pressure. Other reasons include poor patient compliance with taking their drugs.

Combining drugs that lower high blood pressure and have similar ways of working in the body may help high blood pressure and lower the risk for medication-related side effects. One of several drug combinations recommended for the treatment of high blood pressure is an angiotensin receptor blocker and a thiazide diuretic. Guidelines also note that combination tablets may improve patient compliance with taking their drugs.

Candesartan is an angiotensin type-1 receptor blocker. Hydrochlorothiazide is a diuretic with blood pressure-lowering effect. This study will combine both of these drugs in one pill and see how it works in people taking part in this study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of essential hypertension.
* Has Systolic Blood Pressure between 150 mmHg and 200 mmHg AND Diastolic Blood Pressure between 110 mmHg and 120 mmHg.
* Has not received any antihypertensive treatment so far.
* Has a negative pregnancy test at baseline in females of childbearing potential. Male and female participants with reproductive potential must use an approved contraceptive method during study treatment evaluation

Exclusion Criteria:

* Has a known or suspected secondary hypertension or primary hyperaldosteronism.
* Has impaired renal function.
* Has severe hepatic impairment.
* Has bilateral renal artery stenosis, solitary kidney or post-renal transplant status.
* Has a history of myocardial infarction, coronary artery bypass graft, percutaneous coronary intervention or cerebral accident (stroke or transient ischaemic attack) within the last 6 months.
* Has a diagnosis or suspicion of the following conditions: hypertrophic obstructive cardiomyopathy, angina pectoris, chronic heart failure, peripheral arterial occlusive disease, hypertensive retinopathy.
* Has hemodynamically relevant stenosis of the aortic or mitral valve.
* Has clinically relevant and refractory hypokalaemia or hyperkalaemia.
* Has uncorrected volume or sodium depletion.
* Has gout or relevant hyperuricaemia.
* Has a known intolerance/hypersensitivity to Candesartan cilexetil or Hydrochlorothiazide.
* Has a known galactose intolerance, lactase deficiency or glucose-galactose malabsorption.
* Is taking psychotropic medication or is addicted to alcohol or drugs.
* Has participated in another trial of an investigational drug or a medical device within the last 30 days or is currently participating in another trial of an investigational drug or a medical device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Systolic Blood Pressure at Week 9. | Baseline and Week 9.
  The change between Systolic Blood Pressure (SBP) value collected at week 9 or final visit and SBP value collected at baseline
Change from Baseline in Diastolic Blood Pressure at Week 9. | Baseline and Week 9.
  The change between Diastolic Blood Pressure (DBP) value collected at week 9 or final visit and DBP value collected at baseline.

SECONDARY OUTCOMES:
Percentage of subjects showing a decrease in SBP to less than 140 mmHg and/or a decrease of SBP by at least 20 mmHg AND a decrease in DBP to less than 90 mmHg and/or a decrease of DBP by at least 10 mmHg. | Week 9.
  Percentage of participants at week 9 or final visit showing a decrease in SBP to less than 140 mmHg and/or a decrease of SBP by at least 20 mmHg AND a decrease in DBP to less than 90 mmHg and/or a decrease of DBP by at least 10 mmHg.
Percentage of subjects showing a decrease in SBP to less than 130 mmHg and/or a decrease of SBP by at least 20 mmHg AND a decrease in DBP to less than 80 mmHg and/or a decrease of DBP by at least 10 mmHg. | Week 9.
  Percentage of participants at week 9 or final visit showing a decrease in SBP to less than 130 mmHg and/or a decrease of SBP by at least 20 mmHg AND a decrease in DBP to less than 80 mmHg and/or a decrease of DBP by at least 10 mmHg.
Change from Baseline in Pulse Rate at Week 9. | Baseline and Week 9.
  The change between Pulse Rate measured at week 9 and Pulse Rate measured at baseline.
Change from Baseline in Systolic Blood Pressure at Final Visit. | Baseline and Final Visit (up to Week 9)
  The change between the Systolic Blood Pressure value collected at week 9 or final visit and the Systolic Blood Pressure value collected at baseline.
Change in Baseline in Diastolic Blood Pressure at Final Visit. | Baseline and Final Visit (up to Week 9)
  The change between the Diastolic Blood Pressure value collected at week 9 or final visit and the Diastolic Blood Pressure value collected at baseline.
Change from Baseline in Pulse Rate at Final Visit. | Baseline and Final Visit (up to Week 9)
  The change between Pulse Rate measured at week 9 or final visit and the Pulse Rate measured at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda Pharma GmbH (Germany)
Locations (16):
- Germany (12):
  - Berlin
  - Blankenhain
  - Dortmund
  - Hamburg
  - Köthen
  - Löhne
  - Nuremberg
  - Remscheid
  - Rodgau
  - Stockach
  - Wardenburg
  - Weinheim
- Ukraine (4):
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Lviv